CLINICAL TRIAL: NCT01703091
Title: A Randomized, Double-Blind, Phase 2 Study of Docetaxel and Ramucirumab Versus Docetaxel and Placebo in the Treatment of Stage IV Non-Small Cell Lung Cancer Following Disease Progression After One Prior Platinum-Based Therapy
Brief Title: A Study of Docetaxel and Ramucirumab Versus Docetaxel and Placebo in the Treatment of Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14658; I4T-JE-JVCG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramucirumab plus Docetaxel (Experimental): Ramucirumab 10 milligram per kilogram (mg/kg) on Day 1 of every 21 day cycle, administered as an intravenous (IV) infusion over approximately 60 minutes. Docetaxel 60 milligram per square meter (mg/m2) on Day 1 of every 21 day cycle, administered as an IV infusion over approximately 60 minutes.
  Interventions: Drug: Ramucirumab; Drug: Docetaxel
- Placebo plus Docetaxel (Placebo Comparator): Placebo (administered at a volume equivalent to a dose of milligram per kilogram (mg/kg)) on Day 1 of every 21 day cycle, administered as an IV infusion over approximately 60 minutes. Docetaxel 60 mg/m2 on Day 1 of every 21 day cycle, administered as an IV infusion over approximately 60 minutes.
  Interventions: Drug: Placebo; Drug: Docetaxel

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY 3009806; IMC-1121B; Cyramza®
  Arms: Ramucirumab plus Docetaxel
Drug: Placebo — Administered IV
  Arms: Placebo plus Docetaxel
Drug: Docetaxel — Administered IV

SUMMARY:
The purpose of this study is to evaluate the effects of ramucirumab in combination with docetaxel in participants with Stage IV non-small cell lung cancer who have had disease progression during or after one prior first-line platinum-based chemotherapy with or without maintenance therapy for advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell Lung Cancer disease
* Clinical stage IV or recurrent disease
* One prior first-line platinum-based chemotherapy regimen with or without maintenance therapy
* For Non-Small Cell Lung Cancer (NSCLC) tumors other than squamous cell histology, the epidermal growth factor receptor (EGFR) mutation status is known prior to randomization
* For participants with activating epidermal growth factor receptor (EGFR) mutation only, prior epidermal growth factor receptor- tyrosine kinase inhibitor (EGFR-TKI) monotherapy (only one regimen in the setting of single use) should be utilized
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version RECIST version 1.1
* Adequate organ function
* Estimated life expectancy of at least 3 months.

Exclusion Criteria:

* Have undergone major surgery within 28 days prior to randomization or have planned major surgery during study treatment
* Receiving concurrent treatment with other anticancer therapy
* Central nervous system disease other than stable and treated brain metastasis
* Has major blood vessel invasion or encasement by cancer
* Has intratumor cavitation
* Has a history of uncontrolled thrombotic disorder
* Is receiving therapeutic anticoagulation with drugs
* Is receiving chronic therapy with nonsteroidal anti-inflammatory drugs
* Has a history of hemoptysis within 2 months prior to randomization
* Has clinically relevant congestive heart failure
* Has experienced any arterial thromboembolic event
* Has uncontrolled arterial hypertension
* Has had a serious or nonhealing wound or, ulcer
* Has significant existing conditions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Japan (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Yoh K, Hosomi Y, Kasahara K, Yamada K, Takahashi T, Yamamoto N, Nishio M, Ohe Y, Koue T, Nakamura T, Enatsu S, Lee P, Ferry D, Tamura T, Nakagawa K. A randomized, double-blind, phase II study of ramucirumab plus docetaxel vs placebo plus docetaxel in Japanese patients with stage IV non-small cell lung cancer after disease progression on platinum-based therapy. Lung Cancer. 2016 Sep;99:186-93. doi: 10.1016/j.lungcan.2016.07.019. Epub 2016 Jul 18. PMID 27565938

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completion was defined as death due to any cause or disease progression.
Groups:
- Ramucirumab Plus Docetaxel: Ramucirumab 10 milligrams/kilogram (mg/kg) administered as an intravenous (IV) infusion over approximately 60 minutes on Day 1 of every 21-day cycle. Docetaxel 60 milligrams/square meter (mg/m2) administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle.
- Placebo Plus Docetaxel: Placebo administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle. Docetaxel 60 mg/m2 administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle.
Period: Overall Study
Arm/Group | Ramucirumab Plus Docetaxel | Placebo Plus Docetaxel
Started | 98 | 99
Received at Least One Dose of Study Drug | 94 | 98
Completed | 89 | 95
Not Completed | 9 | 4
Not completed — Adverse Event | 5 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who had received at least one dose of study drug.
Groups:
- Ramucirumab + Docetaxel: Ramucirumab 10 mg/kg administered as an intravenous (IV) infusion over approximately 60 minutes on Day 1 of every 21-day cycle. Docetaxel 60 mg/m2 administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle.
- Placebo + Docetaxel: Placebo administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle. Docetaxel 60 mg/m2 administered as an IV infusion over approximately 60 minutes on Day 1 of every 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 94 | 98 | 192
Age, Continuous [Median (Full Range); unit: Years] | 63.9 [29 to 78] | 64.1 [27 to 79] | 64 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 66 | 71 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 94 | 98 | 192
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Japan | 94 | 98 | 192

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from baseline until measured progressive disease (PD) or death from any cause, whichever is first. According to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), PD was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the 20% relative increase, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression. Participants without objectively determined PD, who were alive at the end of the follow-up period (or lost to follow-up), were censored on the date of the participant's last complete radiographic tumor assessment; if no baseline or post-baseline radiologic assessment was available, the participant was censored at the date of randomization.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (Up to 21 Months)
Population: Full Analysis Set (FAS) population: All randomized participants who received at least one dose of study drug and whose prior therapy did not include EGFR-TKI monotherapy. The number of censored participant data for ramucirumab and placebo is 13 and 9, respectively.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Months | 5.22 [3.52 to 6.97] | 4.21 [2.83 to 5.62]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from baseline to the date of death from any cause. Participants who were alive at the end of the follow-up period (or lost to follow-up) were censored on the last date the participant was known to be alive.
Time Frame: Baseline to Death from Any Cause (Up to 28 Months)
Population: FAS population: All randomized participants who received at least one dose of study drug and whose prior therapy did not include EGFR-TKI monotherapy. The number of censored participant data for ramucirumab and placebo is 36 and 35, respectively.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Months | 15.15 [12.45 to 26.55] | 14.65 [11.93 to 24.44]

3. Secondary Outcome: Percentage of Participants Who Achieved Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) [Objective Tumor Response Rate (ORR)]
Description: Participants achieved an objective response if they had a best overall response of complete response (CR) or partial response (PR). According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal [ULN]); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. The percentage of participants who achieved an objective response equals (number of participants with CR or PR)/(number of participants assessed)*100.
Time Frame: Baseline to Measured Progressive Disease or Participant Stops Study (Up to 97 Weeks)
Population: FAS population: All randomized participants who received at least one dose of study drug and whose prior therapy did not include EGFR-TKI monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Percentage of Participants | 28.9 [19.1 to 40.5] | 18.5 [10.8 to 28.7]

4. Secondary Outcome: Percentage of Participants Who Achieved Best Overall Disease Response of CR, PR or Stable Disease (SD) [Disease Control Rate (DCR)]
Description: Participants achieved disease control if they had a best overall response of PR, CR or SD. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal [ULN]); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. The percentage of participants who achieved disease control equals (number of participants with CR, PR, or SD)/(number of participants assessed)*100.
Time Frame: Baseline to Measured Progressive Disease or Participant Stopped Study (Up to 97 Weeks)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Percentage of Participants | 78.9 [68.1 to 87.5] | 70.4 [59.2 to 80.0]

5. Secondary Outcome: Change From Baseline in European Quality of Life Questionnaire - 5 Dimension (EQ-5D) Index Score
Description: The EQ-5D is a quality-of-life instrument which allowed participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a scale from 1 to 3 (no problem, some problems, and extreme problems, respectively). These combinations of attributes were converted into a weighted Health State Index score according to a United Kingdom population-based algorithm; the possible values for the Health State Index score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension).
Time Frame: Baseline, Day 21 Each Cycle (Cycle = 21 Days) and 30-Day Follow Up (Up to 97 Weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Units on a Scale
  Cycle 1 (n = 69, 77) | -0.024 (0.1928) | -0.007 (0.1918)
  Cycle 2 (n = 62, 66) | -0.021 (0.2190) | 0.006 (0.1961)
  Cycle 3 (n = 48, 53) | -0.010 (0.2324) | -0.005 (0.1891)
  Cycle 4 (n = 40, 48) | 0.015 (0.1683) | -0.026 (0.1610)
  Cycle 5 (n = 32, 40) | 0.000 (0.2280) | -0.012 (0.1433)
  Cycle 6 (n = 28, 36) | 0.035 (0.1741) | -0.005 (0.1409)
  Cycle 7 (n = 25 ,31) | 0.002 (0.1857) | -0.039 (0.1282)
  Cycle 8 (n = 23, 30) | -0.053 (0.1750) | -0.071 (0.1800)
  30-Day Follow Up (n= 56, 70) | -0.102 (0.2209) | -0.132 (0.3344)

6. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scale (LCSS)
Description: The participant-reported LCSS was a 9-item questionnaire. Six items were symptom-specific measures for lung cancer (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain), and 3 summation items described total symptomatic distress, interference with activity level, and global quality of life. Participant responses to each item were measured using a visual analog scale (VAS) from 0 (best outcome) to 100 (worst outcome). The Average Symptom Burden Index (ASBI) was the mean of the 6 symptom-specific items in the LCSS. The Total LCSS was the mean of all 9 LCSS items. Maximum improvement in LCSS scores, ASBI, and Total LCSS score was the largest decrease from baseline for each variable, which was the smallest (most negative or smallest positive) non-missing value among all change from baseline values for each variable.
Time Frame: Baseline to Measured Progressive Disease or Participant Stopped Study (up to 97 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 76 | 81
Millimeter
  Loss of Appetite (n=73, 79) | -12.5 (26.23) | -16.2 (21.45)
  Fatigue (n=73, 80) | -4.9 (25.38) | -7.8 (23.59)
  Cough (n=73, 80) | -4.4 (23.10) | -18.3 (23.83)
  Dyspnea (n=73, 80) | -4.7 (23.09) | -8.7 (20.16)
  Hemoptysis (n=73, 80) | -1.2 (12.83) | -3.7 (17.25)
  Pain (n=73, 80) | -9.6 (23.66) | -9.0 (21.52)
  Overall Symptoms (n=73, 80) | -7.1 (26.10) | -11.5 (19.83)
  Interference with Activity Level (n=73, 80) | -8.4 (25.84) | -11.9 (21.98)
  Quality of Life (n=73, 80) | -11.7 (28.06) | -12.7 (21.06)
  ASBI (n=73, 79) | -2.82 (14.93) | -6.93 (12.06)
  Total LCSS (n=73, 79) | -3.20 (15.64) | -7.13 (11.74)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Serious Adverse Events (participants affected / at risk) | 30/94 | 31/98
Other Adverse Events (participants affected / at risk) | 94/94 | 98/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Docetaxel (N=94) | Placebo + Docetaxel (N=98)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 6 (6)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Docetaxel (N=94) | Placebo + Docetaxel (N=98)
Anaemia (Blood and lymphatic system disorders) | 37 (60) | 41 (68)
Febrile neutropenia (Blood and lymphatic system disorders) | 26 (29) | 15 (17)
Leukopenia (Blood and lymphatic system disorders) | 13 (33) | 24 (63)
Neutropenia (Blood and lymphatic system disorders) | 17 (46) | 30 (70)
Eye discharge (Eye disorders) | 5 (5) | 1 (1)
Lacrimation increased (Eye disorders) | 8 (8) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 15 (34) | 28 (36)
Diarrhoea (Gastrointestinal disorders) | 31 (50) | 23 (50)
Nausea (Gastrointestinal disorders) | 34 (52) | 39 (52)
Periodontal disease (Gastrointestinal disorders) | 6 (7) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 50 (92) | 31 (41)
Vomiting (Gastrointestinal disorders) | 14 (15) | 22 (31)
Face oedema (General disorders) | 15 (18) | 7 (7)
Fatigue (General disorders) | 29 (45) | 25 (47)
Malaise (General disorders) | 43 (97) | 47 (85)
Oedema peripheral (General disorders) | 34 (38) | 28 (33)
Pyrexia (General disorders) | 31 (54) | 26 (45)
Hypersensitivity (Immune system disorders) | 3 (3) | 5 (15)
Conjunctivitis (Infections and infestations) | 6 (6) | 2 (2)
Lung infection (Infections and infestations) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (9) | 11 (11)
Paronychia (Infections and infestations) | 6 (6) | 7 (7)
Pharyngitis (Infections and infestations) | 8 (9) | 2 (2)
Skin infection (Infections and infestations) | 5 (5) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 9 (14) | 5 (7)
Alanine aminotransferase increased (Investigations) | 15 (17) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 19 (26) | 6 (12)
Blood bilirubin increased (Investigations) | 3 (4) | 6 (11)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (16) | 11 (43)
Neutrophil count decreased (Investigations) | 73 (281) | 69 (219)
Platelet count decreased (Investigations) | 22 (42) | 14 (22)
Weight decreased (Investigations) | 5 (6) | 9 (12)
White blood cell count decreased (Investigations) | 73 (261) | 68 (226)
Decreased appetite (Metabolism and nutrition disorders) | 54 (90) | 51 (92)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 29 (44) | 21 (32)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (24) | 14 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 13 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (32) | 18 (26)
Dizziness (Nervous system disorders) | 4 (4) | 6 (7)
Dysgeusia (Nervous system disorders) | 25 (36) | 26 (34)
Headache (Nervous system disorders) | 12 (16) | 16 (22)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (20) | 27 (27)
Insomnia (Psychiatric disorders) | 17 (18) | 18 (21)
Proteinuria (Renal and urinary disorders) | 28 (36) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 46 (90) | 18 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 (24) | 9 (24)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 63 (63) | 61 (62)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 (9) | 12 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (18) | 17 (17)
Nail discolouration (Skin and subcutaneous tissue disorders) | 22 (22) | 19 (19)
Nail ridging (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Onychomadesis (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (11) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 12 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (8)
Flushing (Vascular disorders) | 4 (12) | 7 (12)
Hypertension (Vascular disorders) | 10 (10) | 0 (0)
Vasculitis (Vascular disorders) | 2 (2) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days